CLINICAL TRIAL: NCT01266031
Title: Phase I/II Adaptive Randomized Trial of Bevacizumab Versus Bevacizumab Plus Vorinostat in Adults With Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: M.D. Anderson Cancer Center (Other); Genentech, Inc. (Industry); Merck Sharp & Dohme LLC (Industry); Brain Tumor Trials Collaborative (Other); Ohio State University (Other); Northwestern University Feinberg School of Medicine (Other); UF Health Cancer Center at Orlando Health (Unknown); Baylor Health Care System (Other); MUSC Hollings Cancer Center (Unknown); University of Utah Health System (Unknown); University of Washington (Other); Henry Ford Health System (Other); Columbia University (Other); Rush University Medical Center (Other); Endeavor Health (Other); The Cleveland Clinic (Other); University of North Carolina, Chapel Hill (Other); Washington University School of Medicine (Other); Texas Oncology-Austin (Unknown)
Responsible Party: Principal Investigator, Mark Gilbert, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999916116; 16-C-N116
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Malignant Glioma; Recurrent Glioblastoma
Keywords: Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Vorinostat; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bevacizumab (Experimental): 10 mg/kg/dose by vein on days 1 and 15 of a 28 day cycle.
  Interventions: Drug: bevacizumab
- Vorinostat and Bevacizumab (Experimental): Vorinostat: 400 mg/day by mouth on days 1 to 7 and days 15 to 21 of a 28 day cycle.
  Bevacizumab: 10 mg/kg/dose by vein on days 1 and 15 of a 28 day cycle.
  Interventions: Drug: vorinostat; Drug: bevacizumab

INTERVENTIONS:
Drug: vorinostat — Vorinostat 400mg/day will be administered on day 1 to 7 and day 15 to 21 orally on a 28 day cycle in the arm with combination of vorinostat and bevacizumab. Vorinostat will be administered orally. Vorinostat capsules should not be opened or crushed and must be administered whole.
  Other Names: Zolinza
  Arms: Vorinostat and Bevacizumab
Drug: bevacizumab — Bevacizumab 10mg/kg will be administered on day 1 and 15 intravenously on a 28 day cycle in both arms.
  Other Names: Avastin

SUMMARY:
The goal of this Phase I portion of this clinical research study is to find the highest tolerable dose of bevacizumab with or without vorinostat, that can be given to patients with malignant gliomas. The safety of these drug combinations will also be studied.

The goal of this Phase II part of this clinical research study is to learn if bevacizumab when given with or without vorinostat can help to control malignant gliomas. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
Background

* Glioblastoma (GBM) is the most common primary brain tumor. With optimal treatment, consisting of focal radiotherapy with concurrent chemotherapy, followed by adjuvant chemotherapy, median survival is 14.6 months. Most patients have evidence of tumor progression within one year of diagnosis despite treatment. At progression, treatment options are limited and mostly ineffective.
* Given the importance of angiogenesis in GBM, anti-angiogenic therapy is a promising strategy in recurrent GBM. Bevacizumab, the first angiogenesis inhibitor approved against cancer by FDA based on improved survival of advanced colon cancer patient, has recently been studied in the GBM.
* The present study aims to determine the potential of vorinostat, an HDAC inhibitor plus bevacizumab, versus bevacizumab alone, in an attempt to increase the anti-angiogenic effects of VEGF by blocking the evasive resistance by combination with vorinostat and to also not only provide the potential of the independent effects of both agents but also the potential for synergy.

Objectives

* To determine the maximum tolerated dose (MTD) of vorinostat plus bevacizumab in adult patients with malignant glioma.
* To determine the efficacy of vorinostat plus bevacizumab versus bevacizumab alone in patients with recurrent WHO grade IV glioma (glioblastoma and gliosarcoma) as determined by progression free survival (PFS) using an adaptive randomization phase II trial design.

Eligibility

* Patients must have histologically proven glioblastoma, gliosarcoma or anaplastic glioma to be eligible for the Phase I component of this protocol. Anaplastic gliomas include anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant glioma NOS (not otherwise specified). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a malignant glioma is made. Only patients with histologically proven or imaging proven recurrent glioblastoma or gliosarcoma will be eligible for the Phase II component.
* Patients must have shown unequivocal evidence for tumor progression as determined by an MRI scan done prior to study entry which will be reviewed by the treating physician to confirm and document recurrence.
* No prior treatment with bevacizumab or Vorinostat

Design

The phase I component will assess the MTD of Vorinostat in combination with Bevacizumab. A conventional phase I design will be used and the MTD will be selected using a 3+3 accrual design at each dose level until MTD is determined. A maximum of 18 patients will be recruited to this component of the study.

The phase II component of the trial compares Bevacizumab to Vorinostat+ Bevacizumab in patients with recurrent GBM. The primary outcome is progression free survival. Patients will be randomized between the two arms using a Bayesian adaptive algorithm. Patients will be randomized fairly between the two arms at the start of the trial (for the first 20 patients). Thereafter, as the trial progresses and data accrue, the randomization will become unbalanced in favor of the treatment that, on average, has better results in terms of failure time. Therefore, each successive patient is more likely to receive the treatment with better results, on average. A minimum of 20 and a maximum of 90 patients will be accrued.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be included in the study based on the following criteria.

* Patients must have histologically proven glioblastoma, gliosarcoma or anaplastic glioma to be eligible for the Phase I component of this protocol. Anaplastic gliomas include anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant glioma NOS (not otherwise specified). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a malignant glioma is made. Only patients with histologically proven or imaging proven recurrent glioblastoma or gliosarcoma will be eligible for the Phase II component. Wafer acceptable if recurrence is confirmed.
* All patients must sign an informed consent indicating their awareness of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
* Patients must be 18 years old or older.
* Patients must have a Karnofsky performance status (KPS) equal or greater than 60
* At the time of registration:

  * Patients must have recovered from the toxic effects of prior therapy to < grade 2 toxicity per CTC version 4 (except deep vein thrombosis )

    1. 28 days from any investigational agent,
    2. 4 weeks (28 days) from prior cytotoxic therapy,
    3. 2 weeks (14 days) from vincristine,
    4. 6 weeks (42 days) from nitrosoureas,
    5. 3 weeks (21 days) from procarbazine administration,
    6. greater than or equal to1 week (7 days) for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count).
* Patients who receive anticancer agents for non-therapeutic purposes unrelated to this study (such as presurgically for obtaining pharmacology data for the agent) will be eligible to enter the study provided they have recovered from the toxic effects of the agent if any. Any questions related to the definition of noncytotoxic agents should be directed to the Study Chair.
* Patients must have adequate bone marrow function (ANC greater than or equal to 1,500/mm3, platelet count of greater than or equal to 100,000/mm3), adequate liver function (SGPT less than or equal to 3 times upper limit normal and alkaline phosphatase less than or equal to 2 times upper limit normal, total bilirubin less than or equal to 1.5mg/dl, Patients with high bilirubin levels related to known diagnosis of benign hyperbilirubinemia (Gilbert s syndrome) will be eligible ., and adequate renal function (BUN less than or equal to 1.5 times institutional normal and Creatinine < 1.5 mg/dl) prior to registration. These tests must be performed within 14 days prior to registration.
* Patients must have shown unequivocal evidence for tumor progression as determined by an MRI scan done prior to study entry which will be reviewed by the treating physician to confirm and document recurrence.

Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis using the local institutional standards for such determination including advanced imaging or surgery.

* The baseline on-study MRI scan should be performed within 14 days (+ 3 working days) prior to registration but before starting treatment and on a steroid dose that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and registration (or at that time), a new baseline MRI is required. The same type of scan, i.e., MRI must be used throughout the period of protocol treatment for tumor measurement.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  1. At least 4 weeks (28 days ) have elapsed from the date of surgery and the patients have recovered from the effects of surgery.
  2. Evaluable or measureable disease following resection of recurrent Malignant Glioma is not mandated for eligibility into the study.
  3. To best assess the extent of residual disease post-operatively, a MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required on a stable steroid dosage for at least 5 days.
* Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 12 weeks (84 days) from the completion of radiation therapy to study entry except if there is unequivocal evidence for tumor recurrence (such as histological confirmation or advanced imaging data such as PET scan) in which case at least 4 weeks (28 days) from completion of radiation therapy will suffice.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, MR spectroscopy or surgical/pathological documentation of disease.
* Women of childbearing potential must have a negative B-HCG pregnancy test documented within 14 days prior to registration. Women of childbearing potential must not be pregnant, must not be breast-feeding, and must practice adequate contraception for the duration of the study, and for 30 days after the last dose of study medication. Patients must not be pregnant because animal studies show that bevacizumab and Vorinostat are teratogenic.
* Male patients on treatment with Vorinostat must agree to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication.
* Patient must be able to tolerate the procedures required in this study including periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study.
* Patients receiving treatment with any antiepileptic medications except Valproic acid (because of its HDAC inhibitory activity) can be included in the study. Vorinostat is not metabolized by Cytochrome P450 3A4 (CYP 3A4); however, Vorinostat may potentially suppress CYP 3A4 activity. Therefore, patients should preferably be treated with nonenzyme inducing anti-epileptic medications although this is not mandatory. If enzyme inducing antiepileptic drugs are used, monitoring of these drug levels should be considered, as considered clinically appropriate by the treating physician.
* For the Phase II portion of the study, patients may have had treatment for no more than 2 prior relapses. There is no limit to the number of relapses for the phase I portion of the study provided the functional status and other eligibility criteria for enrollment are met. Relapse is defined as progression following initial therapy (i.e. radiation+/- chemo if that was used as initial therapy). The intent therefore is that patients had no more than 3 prior therapies (initial and treatment for 2 relapses). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse. For patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse

EXCLUSION CRITERIA:

General Exclusion Criteria

* Inability to comply with protocol or study procedures (for example, an inability to swallow tablets).
* Prior treatment with bevacizumab or Vorinostat.
* Patients receiving valproic acid (VPA), an anticonvulsant drug with HDAC inhibitor properties, will be excluded, unless they are switched to an alternative agent prior to treatment initiation. A 5-day wash out period is required. Patients who have failed prior treatment with other histone deacetylase inhibitors will be excluded.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent.
* Any condition, including the presence of clinically significant laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study. These would include

  1. Active infection (including persistent fever) including known AIDS or Hepatitis C infection
  2. Diseases or conditions that obscure toxicity or dangerously alter drug metabolism
  3. Serious intercurrent medical illness (e.g. symptomatic congestive heart failure).
* Current, recent (within 4 weeks (28 days) of the first infusion of this study, or planned participation in an experimental antitumor drug study (other than the current one).
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix or bladder), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients with spinal disease (metastasis) and/or leptomeningeal disease will not be allowed in the study.

Bevacizumab-Specific Exclusion Criteria

* Inadequately controlled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg).
* Prior history of hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or unstable angina within 6 months prior to Day 1.
* History of stroke or transient ischemic attack within 6 months prior to Day1.
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1.
* History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study. Patients with recent resection will be eligible for entry into the surgical arm of the study but will follow guidelines as in section 4.9 .
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1.
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1.
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* Proteinuria as demonstrated by:

  * Urine protein: creatinine (UPC) ratio greater than or equal to 1.0 at screening OR
  * Urine dipstick for proteinuria greater than or equal to 2+ (patients discovered to have greater than or equal to 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate less than or equal to 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab.
* Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential is required for study treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-07-12 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Gilbert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: the study was initially written in 2010 and eventually activated at the lead site on 7/6/2011.
Groups:
- Vorinostat + Bevacizumab: Phase I Vorinostat starting dose 400 mg orally days 1 - 7 & days 15 - 21 in combination with Bevacizumab fixed dose 10mg/kg IV on Days 1 & 15 of 28 day cycle.
- Bevacizumab: Phase II Bevacizumab 10 mg/kg/dose IV on days 1 & 15 of a 28 day cycle.
- Bevacizumab + Vorinostat 400 mg: Phase II Bevacizumab 10 mg/kg/dose IV Day 1 & 15 + MTD of Vorinostat 400 mg/day by mouth on days 1 to 7 & days 15 to 21 of a 28 day cycle.
Period: Overall Study
Arm/Group | Vorinostat + Bevacizumab | Bevacizumab | Bevacizumab + Vorinostat 400 mg
Started | 6 | 41 | 49
Completed | 6 | 38 | 47
Not Completed | 0 | 3 | 2
Not completed — Not treated | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat + Bevacizumab: Phase I Vorinostat starting dose 400 mg orally days 1 - 7 and days 15 - 21 in combination with Bevacizumab fixed dose 10mg/kg IV on Days 1 + 15 of 28 day cycle.
- Bevacizumab: Phase II Bevacizumab 10 mg/kg/dose by vein on days 1 and 15 of a 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Vorinostat + Bevacizumab | Bevacizumab | Bevacizumab + Vorinostat 400 mg | Total
Number analyzed (Participants) | 6 | 41 | 49 | 96
Age, Continuous [Median (Full Range); unit: years] | 51.5 [18 to 66] | 60 [27 to 88] | 57 [22 to 75] | 57 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 18 | 33
  Male | 3 | 29 | 31 | 63
Region of Enrollment [Number; unit: participants]
  United States | 6 | 41 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 6 Months
Description: PFS is time measured in months to disease progression as assessed at six months from participant registration. Assessments continue every 8 weeks up to 28 days after last dose (follow-up), anticipated trial length one year.
  Participants must be assessed at least 4 weeks after surgery to begin treatment in the adaptive randomized Phase 2 portion of the trial. PFS in participants in the surgical arm determined from the date of randomization to the treatment arms and not from the date of registration in the trial.
  Study outcome measure period ended June 2015.
Time Frame: Baseline until disease progression or death due to any cause, up to six months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab | Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 38 | 47
Months | 0.29 [0.15 to 0.45] | 0.23 [0.12 to 0.36]
Statistical Analysis 1: Comparison: Bevacizumab vs Bevacizumab + Vorinostat 400 mg; Null hypothesis is: progression free survival (PFS) 6 months of Bevacizumab = PFS 6 months of Bevacizumab + Vorinostat; Test type: Superiority or Other; p = 0.26, Chi-squared — Null hypothesis is: PFS 6 months of Bevacizumab = PFS 6 months of Bevacizumab + Vorinostat

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Oral Vorinostat Used With Bevacizumab
Description: MTD defined as the dose level at which 1/6 patients experience dose limiting toxicity (DLT), using conventional Phase I design where the MTD was selected using a 3+3 accrual design at each dose level until MTD was determined. Toxicities will be graded according to the Common Terminology Criteria for Adverse events (CTCAE) Version 4.0.
Time Frame: 28 day, cycle 1
Measure: Number; unit: mg/day
Arm/Group | Vorinostat + Bevacizumab
Number analyzed (Participants) | 6
mg/day | 400

3. Secondary Outcome: Time to Progression (TTP)
Description: Progression defined by the Modified MacDonald criteria is 25% increase in the sum of products, of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any lesion/site, OR failure to return for evaluation due to health or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 3, 6, and 12 months from patient registration
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase II: Bevacizumab: Phase II Bevacizumab 10 mg/kg/dose IV on days 1 & 15 of a 28 day cycle.
- Phase II: Bevacizumab + Vorinostat 400 mg: Phase II Bevacizumab 10 mg/kg/dose IV Day 1 & 15 + MTD of Vorinostat 400 mg/day by mouth on days 1 to 7 & days 15 to 21 of a 28 day cycle.
Arm/Group | Phase II: Bevacizumab | Phase II: Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 38 | 47
Months
  Overall TTP | 4.07 [1.94 to 5.88] | 3.71 [2.73 to 4.63]
  3 months | 0.59 [0.41 to 0.73] | 0.62 [0.46 to 0.74]
  6 months | 0.29 [0.15 to 0.45] | 0.28 [0.15 to 0.42]
  12 months | 0.06 [0.01 to 0.19] | 0.15 [0.06 to 0.29]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was computed using the number of months from the date of randomization to the date of death, up to 30 months. Participants still alive were censored at the last follow-up date.
Time Frame: up to 30 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab | Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 38 | 47
Months | 9.24 [5.88 to 11.40] | 7.80 [5.04 to 9.12]

5. Secondary Outcome: Effects of Bevacizumab With and Without Vorinostat Upon Biomarkers of Angiogenesis Vascular Endothelial Growth Factor (VEGF), Placental Growth Factor (PIGF), and Basic Fibroblast Growth Factor (bFGF)
Description: About 5cc of blood was collected to measure plasma angiogenic proteins vascular endothelial growth factor (VEGF), placental growth factor (PIGF), and basic fibroblast growth factor (bFGF) by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline before treatment, Cycle 1 Day 2, day 15 (pre-infusion and post-infusion), Cycle 2 (pre-infusion)
Population: This outcome measure was not done. A few samples were collected and stored. However, the correlative biology was predicated on adequate acquisition of tumor tissue and funding. unfortunately, we were unable to obtain funding to perform this aspect (i.e. analysis) of the study.
Groups:
- Phase I: Vorinostat + Bevacizumab: Phase I Vorinostat starting dose 400 mg orally days 1 - 7 & days 15 - 21 in combination with Bevacizumab fixed dose 10mg/kg IV on Days 1 & 15 of 28 day cycle.
Arm/Group | Phase I: Vorinostat + Bevacizumab | Phase II: Bevacizumab | Phase II: Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Effects of Bevacizumab With and Without Vorinostat Upon Biomarkers of Angiogenesis Stromal Cell-derived Factor α (SDF1α), and Angiopoietin 1 (Ang 1) and 2 (Ang 2) by Enzyme-linked Immunosorbent Assay (ELISA)
Description: About 5cc of blood was collected to measure plasma angiogenic proteins stromal cell-derived factor α (SDF1α), angiopoietin 1 and 2 by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline before treatment, Cycle 1 Day 2, day 15 (pre-infusion and post-infusion), Cycle 2 (pre-infusion)
Population: as for outcome 5
Arm/Group | Vorinostat + Bevacizumab | Bevacizumab | Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Patients Rating Their Symptoms to be 7 or Greater on a 0-10 Scale Using the Mean Severity of the MD Anderson Symptom Inventory-Brain Tumor Module (MDSAI-BT) Self Reporting Tool
Description: Percentage of patients rating their symptoms to be 7 or greater on a 0-10 scale using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) Self Reporting Tool. Zero is "not present" and 10 is "as bad as you can imagine. All patients with at least one valid questionnaire will be included in the analyses. Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom severity and symptom interference measures.
Time Frame: Baseline, week 4, week 8, and end of therapy, approximately week 52 (cycle 12)
Population: Reason outcome measure #7 is not done per arm/group is it was intentionally not completed due to negative findings of the study's primary outcomes.
Measure: Number; unit: percentage of of participants
Groups:
- All Participants: All participants who received at least one dose of Bevacizumab by vein and/or Bevacizumab (by vein) + Vorinostat by mouth of a 28 day cycle.
Arm/Group | All Participants
Number analyzed (Participants) | 50
percentage of of participants
  Baseline | 2
  Cycle 2, week 4: number analyzed (Participants) | 31
  Cycle 2, week 4 | 0
  Cycle 4, week 8: number analyzed (Participants) | 21
  Cycle 4, week 8 | 0
  End ot therapy, week 52: number analyzed (Participants) | 28
  End ot therapy, week 52 | 0

8. Secondary Outcome: Mean Symptom Severity Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) Self Reporting Tool
Description: Overall mean severity of 22 symptoms. Symptoms are rated 0-10, zero is "not present" and 10 is "as bad as you can imagine". All patients with at least one valid questionnaire will be included in the analyses.
Time Frame: Baseline, week 4 (cycle 2), week 8 (cycle 4), and end of therapy, approximately week 52 (cycle 12)
Population: Overall analysis was done but not done by treatment arm/group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 50
score on a scale
  Baseline | 1.6 (1.5)
  Cycle 2: number analyzed (Participants) | 31
  Cycle 2 | 1.3 (1.1)
  Cycle 4: number analyzed (Participants) | 21
  Cycle 4 | 1.9 (1.6)
  End of therapy: number analyzed (Participants) | 28
  End of therapy | 2.2 (1.7)

9. Secondary Outcome: Mean Symptom Interference at the Time of Clinical Evaluation
Description: Overall mean interference severity of 6 interference items. Interference is rated 0-10, zero is "did not interfere" and 10 is "as bad as you can imagine". All patients with at least one valid questionnaire will be included in the analyses.
Time Frame: Baseline, (cycle 2), week 8 (cycle 4), and end of therapy, approximately week 52 (cycle 12)
Population: Overall analysis was done but not done by treatment arm/group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 50
score on a scale
  Baseline | 2.2 (2.4)
  Cycle 2: number analyzed (Participants) | 32
  Cycle 2 | 1.7 (1.7)
  Cycle 4: number analyzed (Participants) | 21
  Cycle 4 | 2.9 (2.4)
  End of therapy: number analyzed (Participants) | 29
  End of therapy | 2.9 (2.6)

10. Secondary Outcome: Radiological Response
Description: Magnetic resonance imaging (MRI) and contrast-enhanced (CE) MRI was used to evaluate tumor response. Response is defined by the Modified MacDonald criteria. Complete Response (CR) is complete disappearance of all measurable and evaluable disease. Partial response (PR) is greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. Partial Response, Non-Measurable (PRNM) is not applicable. Stable/No Response does not qualify for CR, PR or progression. Progression is 25% increase in the sum of products, of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any lesion/site, OR failure to return for evaluation due to health or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: End of therapy, approximately
Population: This outcome measure was not done. We collected radiological response data provided by the local physician at time points per protocol. At the end of the study, the plan was to send all MRI discs to one radiologist for central review to confirm responses. With only limited funding, and negative findings, the PI decided to not pursue this outcome.
Arm/Group | Vorinostat + Bevacizumab | Bevacizumab | Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Phase I adverse events collected within 4 week (28 day) cycle. Phase II evaluated for adverse events after each cycle for first 2 cycles and subsequently after each 2 cycles of treatment prior to initiating the next cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat + Bevacizumab | Bevacizumab | Bevacizumab + Vorinostat 400 mg
Number analyzed (Participants) | 6 | 38 | 47
Participants | 6 | 38 | 47

ADVERSE EVENTS:
Time Frame: Phase I adverse events collected within 4 week (28 day) cycle. Phase II evaluated for adverse events after each cycle for first 2 cycles and subsequently after each 2 cycles of treatment prior to initiating the next cycle.
Description: The summary is based on the information of the 85 treated patients. A total of 1098 adverse events have been observed in 82 patients after they started the treatment.
Arm/Group | Phase I: Vorinostat + Bevacizumab | Phase II: Bevacizumab | Phase II: Bevacizumab + Vorinostat 400 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/38 | 1/47
Serious Adverse Events (participants affected / at risk) | 0/6 | 10/38 | 14/47
Other Adverse Events (participants affected / at risk) | 6/6 | 36/38 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Vorinostat + Bevacizumab (N=6) | Phase II: Bevacizumab (N=38) | Phase II: Bevacizumab + Vorinostat 400 mg (N=47)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 5 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Blood and Lymphatic System Disorders, Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders, Other specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders, Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Vorinostat + Bevacizumab (N=6) | Phase II: Bevacizumab (N=38) | Phase II: Bevacizumab + Vorinostat 400 mg (N=47)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (4)
Ear and labyrinth disorders, Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase (ALT) increased (Investigations) | 2 (4) | 2 (3) | 4 (6)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 3 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 5 (5) | 15 (17)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase (AST) increased (Investigations) | 2 (4) | 1 (2) | 3 (4)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Bicarbonate Serum-low (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1) | 3 (3)
Blurred vision (Eye disorders) | 1 (2) | 2 (3) | 2 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 2 (4)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (2) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 5 (6) | 6 (8)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 3 (5) | 3 (4)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6) | 4 (4) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8) | 5 (6)
Creatinine increased (Investigations) | 1 (1) | 4 (7) | 3 (5)
Cushingoid (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
DECUBITUS Ulcer Sacrum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (4) | 5 (5)
Bump at sutura site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple scabs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 4 (6) | 9 (20)
Diplopia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 3 (4) | 11 (11)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2)
Dysphasia (Nervous system disorders) | 0 (0) | 4 (6) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 6 (6)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 6 (8) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 7 (10)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 5 (6)
Fatigue (General disorders) | 6 (11) | 10 (16) | 22 (31)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 4 (7) | 5 (8) | 4 (5)
Gait/walking (wide based ataxic hemiparetic) (General disorders) | 2 (2) | 0 (0) | 0 (0)
Gait/walking Impaired mobility (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Gastrointestinal (sensitivity to smell) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 2 (4) | 3 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (10) | 11 (14) | 11 (21)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin Increase (Investigations) | 5 (9) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (19) | 10 (17) | 10 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 19 (57) | 18 (41)
Hypertriglycedidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (6) | 4 (5) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (9) | 4 (5) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Infection with Normal ANC (Neck NOS), cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with Normal ANC (Neck NOS), herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with Normal ANC (Neck NOS), (Urinary Tract NOS) (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Infection with Normal ANC (Wound), Herpes Z-back-perineal-scrutum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 6 (6) | 2 (2)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
International normalized ratio (INR) increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (4) | 4 (4)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 1 (1)
Irregular Menses (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 3 (10) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 3 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (24) | 7 (8) | 4 (10)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 4 (5) | 10 (11) | 11 (13)
Mental Status Altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (Elevated BUN) (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (elevated LDH) (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (high chloride) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (low chloride) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (low creatinine) (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (low protein) (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
METABOLIC/LABORATORY (low uric acid) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Mood Alteration (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Muscle weakness- Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness lower extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 7 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 2 (3)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8) | 6 (7) | 16 (20)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (4) | 11 (24)
Neuropathy, Numbness, Right sided (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy, Cranial (Pupil, Upper eyelid) (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0)
Neuropathy, Sensory Legs/Toes tingling (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 8 (16)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Obstruction GI (STOMACH-small bowel nos) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OCULAR SURFACE DISEASE (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OCULAR/VISUAL (Right homonymous hemianopsia) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OCULAR/VISUAL (Right & Left visual field deficits) (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2) | 6 (8)
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (Neuropathic in perineal/buttock) (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 4 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2) | 5 (6)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 5 (5) | 6 (9) | 11 (19)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (4) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Pyramidal Tract Dysfunction (Nervous system disorders) | 4 (8) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 5 (7) | 6 (7)
Sensory loss left side (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (5)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (8) | 3 (4)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4)
Speech Impairment (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Taste Alteration (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (6)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 3 (4) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (6)
Weight gain (Investigations) | 0 (0) | 2 (2) | 3 (4)
Weight loss (Investigations) | 1 (1) | 3 (5) | 6 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (2) | 5 (13)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (6)
Hyperpigmentation (hands & knuckles) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT01266031/Prot_SAP_000.pdf